CLINICAL TRIAL: NCT06845059
Title: The "11 for Health" Program and Its Impact on Physical Fitness, Health Status, Health Knowledge, and Pro-Health Behaviors of Children in Poland
Brief Title: The "11 for Health" Program Intervention and Its Impact on Polish Children
Acronym: 11FHPoland
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Adrian Drożdżowski, MSc, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: WroclawUHSS Ethics (21/2024)
Record Dates: First submitted 2025-02-14; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Health Knowledge; Fitness; Wellbeing; Health Behavior; Attitude
Keywords: FIFA 11 For Health
MeSH Terms: conditions — Health Behavior; Behavior | interventions — Health

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Physical Education (Control group) (No Intervention): Participants will participate in standard physical education (PE) classes with no additional interventions.
- "11 For Health" Program (Intervention group) (Experimental)
  Interventions: Other: "11 For Health"

INTERVENTIONS:
Other: "11 For Health" — Participants will participate in the "11 For Health" program, consisting of 11 sessions over 11 weeks. The program combines football skills with health education to promote overall health and well-being.
  Arms: "11 For Health" Program (Intervention group)

SUMMARY:
This study evaluates the impact of the "11 For Health" program-an innovative football-based health education initiative-on children's physical fitness, health status, health knowledge, and pro-health behaviors. Originally implemented in African and South American countries, the program has been adapted and successfully introduced in European and Asian countries. The intervention consists of structured football sessions integrating health education messages aimed at promoting a healthy lifestyle among schoolchildren. The study aims to evaluate the effectiveness of this program in enhancing both physical fitness and health-related outcomes in comparison to traditional physical education classes

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will include children from schools that have volunteered to participate in the project. These schools will be assigned to clusters, which will then be randomly allocated to one of two groups: the control group, following the standard physical education curriculum, or the intervention group, participating in the "11 For Health" program over an 11-week period (two sessions per week, 45 minutes each). Within each school, all students in a given cluster will be assigned to the same group to ensure consistency and minimize potential contamination.

Structure of the "11 For Health" Program The "11 For Health" programis a football-based program combined with structured health education content which consists of 11 structured sessions, each lasting 90 minutes and divided into two parts: • "Play Football" - A practical football-based component where children engage in skill-building exercises such as passing, dribbling, and shooting. • "Play Fair" - A theoretical component focused on health education, where key health-related topics (e.g., nutrition, hygiene, physical activity) are introduced through interactive discussions and activities.A new football-related topic paired with an appropriate health message will be discussed each week. Each session follows a standardized manual that outlines learning objectives, football exercises, and health messages. The program is designed to foster both physical engagement and health awareness, reinforcing messages through active participation. Children in the intervention group will participate in the "11 For Health" program during their weekly physical education lessons. In the Polish education system, children typically have 180 minutes of physical education per week. Of this, 90 minutes will be dedicated to the "11 For Health" program, while the remaining time will be spent on the standard physical education curriculum. This will allow for a direct comparison of the impacts of the program against the standard curriculum.

Participants will undergo baseline (pre-test) and post-intervention (post-test) assessments to evaluate physical fitness, health-related knowledge, wellbeing, body composition, health status, and pro-health behaviors. Physical tests and questionnaires will be used to measure outcomes. Physical fitness will be assessed using tests evaluating balance, muscular strength, aerobic capacity, agility, and endurance. Body composition will be analyzed through anthropometric measurements and bioelectrical impedance analysis (BIA), while cardiovascular health will be evaluated by measuring resting heart rate and blood pressure. Health-related knowledge, wellbeing, dietary habits, and physical activity levels will be assessed using questionnaires. Following the intervention, children in the experimental group will report their level of enjoyment of the program and football in general using a 5-point Likert scale. Teachers will complete questionnaires assessing program feasibility, acceptability, and implementation challenges. After the program's completion and data collection, a comparative analysis of the results from both groups will be conducted to determine the impact of the "11 For Health" program in improving physical fitness, health knowledge, health status, overall well-being and pro-health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Age between 9 and 14 years,
* Signed informed consent from a parent or legal guardian for underage participants.

Exclusion Criteria:

* Disabilities.
* Medical contraindications.
* Medical or other exemptions from physical education classes.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Health Knowledge | Baseline and after 3 months (post-intervention)
  Health knowledge will be assessed using the "11 For Health" Health Knowledge Questionnaire. This questionnaire evaluates children's understanding of key health topics, including nutrition, physical activity, and hygiene. It consists of multiple-choice questions, aimed at measuring the knowledge acquired during the program. Higher scores indicate greater health knowledge (min= 0, max= 36)
Wellbeing | Baseline and after 3 months (post-intervention)
  Wellbeing will be assessed using the Kidscreen-27 questionnaire, which evaluates emotional well-being, social functioning, and general life satisfaction. It uses a Likert scale to assess happiness, relationships with family, and feelings of self-worth, capturing the child's overall perception of their quality of life. Higher scores indicate better well-being. Higher scores indicate better well-being (Minimum = 27, Maximum = 135).
Yo-Yo Intermittent Recovery Test Level 1 (YYIR1C) | Baseline and after 3 months (post-intervention)
  Aerobic fitness and endurance will be assessed using the Yo-Yo Intermittent Recovery Test Level 1 (YYIR1C), which measures the total distance covered in a repeated sprint and recovery format. A greater distance (meters [m]) indicates better aerobic capacity.
Stork Balance Test | Baseline and after 3 months (post-intervention)
  Balance performance will be assessed using the Stork Balance Test, which evaluates single-leg balance ability. Time held in seconds ( higher scores indicate better balance).
Standing Long Jump Test | Baseline and after 3 months (post-intervention)
  Lower body explosive strength will be assessed using the Standing Long Jump Test, measuring the horizontal distance jumped from a standing position with hands positioned on hips. A longer (centimeters [cm]) jump indicates better lower-body power
Hand Grip Test | Baseline and after 3 months (post-intervention)
  Muscular strength will be assessed using the Hand Grip Test, which measures maximal isometric grip strength. Measured in kilograms [kg] (higher values = greater grip strength).
Plank Test | Baseline and after 3 months (post-intervention)
  Core endurance will be assessed using the Plank Test, measuring the duration a participant can hold a plank position. A longer (seconds [s]) duration indicates better core endurance.
20m Sprint Test | Baseline and after 3 months (post-intervention)
  Speed and acceleration will be assessed using the 20m Sprint Test, measuring the time taken to cover a 20-meter distance. A shorter time (seconds [s]) indicates better sprint performance.
Resting Heart Rate | Baseline and after 3 months (post-intervention)
  Cardiovascular health will also be assessed by measuring resting heart rate (HR) using an electronic heart rate monitor. Lower resting heart rate (Beats per minute [bpm]) generally indicates better cardiovascular fitness.
Systolic Blood Pressure | Baseline and after 3 months (post-intervention)
  Cardiovascular health will be assessed by measuring resting systolic blood pressure using an electronic blood pressure monitor. Lower values (Millimeters of mercury [mmHg]) within a normal range indicate better cardiovascular health.
Diastolic blood pressure | Baseline and after 3 months (post-intervention)
  Cardiovascular health will be assessed by measuring resting diastolic blood pressure using an electronic blood pressure monitor. Lower values (millimeters of mercury [mmHg]) within a normal range indicate better cardiovascular health.
Body Fat Percentage | Baseline and after 3 months (post-intervention)
  Body fat percentage will be assessed using an electronic bioimpedance tool (InBody 270) to determine the proportion of body weight composed of fat. Lower values (percentage [%]) within a healthy range indicate better body composition.
Skeletal Muscle Mass | Baseline and after 3 months (post-intervention)
  Skeletal muscle mass will be assessed using an electronic bioimpedance tool (InBody 270) to measure the total mass of skeletal muscles in the body. Higher values (kilograms [kg]) indicate greater muscle mass.

SECONDARY OUTCOMES:
Dietary habits | Baseline and after 3 months (post-intervention)
  Dietary habits will be evaluated using the SF-FFQ4PolishChildren questionnaire. This tool assesses food frequency and dietary choices in children, including the types of foods consumed, frequency of consumption, and general eating habits. Higher scores indicate more frequent consumption of a given food group. The questionnaire assesses dietary quality based on eating habits and food intake frequency.
Physical activity | Baseline and after 3 months (post-intervention)
  Physical activity levels will be assessed using the Modified PAQ-C ( Modified Physical Activity Questionnaire for Children). This questionnaire gathers information on the frequency and intensity of physical activities, including sports, outdoor play, and other forms of exercise. Higher scores indicate greater levels of physical activity.
Programme enjoyment | After 3 months (post-intervention)
  The enjoyment of the "11 For Health" program and football in general will be assessed through questions like "How did you like the '11 For Health' program?" and "How fun do you think football is?" Responses will be recorded on a 5-point Likert scale to measure the child's (intervention group) enjoyment and overall satisfaction with the program. Higher scores (points, [min=2, max=10]) indicate higher enjoyment level.
Body height (BH) | Baseline and after 3 months (post-intervention)
  Body height will be measured from the base to the vertex (top of the head) using a stadiometer to provide accurate data on the child's growth and development.
Body weight (BW) | Baseline and after 3 months (post-intervention)
  Body weight will be measured using an electronic scale (InBody), providing precise data on body weight. This method is commonly used in clinical and research settings.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Chmura, Professor, Study Director — Wroclaw University of Health and Sport Sciences
Locations (1):
- Wroclaw University of Health and Sport Sciences, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) will only be shared in the form of published scientific articles, which will include anonymized results and analyses. Individual-level data will not be shared directly.
Supporting Information: Study Protocol, SAP, CSR